CLINICAL TRIAL: NCT01074736
Title: Host Genetic Susceptibility to Avian Influenza A/H5N1 in Vietnam, Thailand, Indonesia and Singapore
Brief Title: Host Genetic Susceptibility to Avian Influenza A/H5N1
Status: Completed | Type: Observational
Sponsor: South East Asia Infectious Disease Clinical Research Network (Network)
Collaborators: University of Oxford (Other); Wellcome Trust (Other)
Responsible Party: Peter Horby, NCC Oxford University Clinical Research Unit - The Hospital for Tropical Diseases, Vietnam
Other Study IDs: SEA 007
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Influenza A Virus/H5N1 Subtype
Keywords: influenza A/H5N1; host genetic susceptibility; genotyping

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * whole blood in tubes containing EDTA
  * mouth wash.
  * buffy coat; cell pellet from centrifuged blood, nucleic acid extracted for diagnostic purposes, serum, throat, nose or endotracheal swabs
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The identification and characterization of susceptibility loci for H5N1 infection in humans could have profound implications. The detection of host genetic factors may shed light on key pathogenic interactions between H5N1 and human cells, assisting in identifying the viral characteristics determining pandemic potential. In addition, the identification and verification of susceptibility loci would be followed by functional studies which might point the way to new therapeutic and preventive options.

The objective of this study is to investigate if host genetic factors are associated with susceptibility to influenza H5N1 illness

DETAILED DESCRIPTION:
This is primarily an hypothesis screening exercise and while guesses based on biological plausibility are possible, a comprehensive analysis of genetic susceptibility can only be achieved by a whole genome approach. Therefore we will test for genetic linkage and association using a large number of Single Nucleotide Polymorphisms (SNPs) spanning the whole genome.

Principal Investigators have access to information on all surviving and deceased laboratory confirmed H5N1 cases. These cases will form the study base. The epidemiologist will attempt to make telephone contact with either the recovered patient or,if the patient died, the closest relative of the deceased patient. The proposed study will be explained and permission will be sought for the epidemiologist and a study nurse to visit the household to explain the study in greater detail, to offer an opportunity for questions and, if the subject agrees, to obtain informed consent for participation. If the epidemiologist has difficulty in making contact with the case or their family the local public authorities will be asked to assist in making contact. Eligible family members of H5N1 cases will be identified by face-to-face interviews with the surviving confirmed cases or close family members of deceased cases.

ELIGIBILITY:
Inclusion Criteria:

* The individual had a clinically compatible illness (defined as respiratory symptoms and an abnormal chest x-ray or encephalitis), AND
* Influenza A/H5 RNA identified in a clinical sample by reverse transcription-polymerase chain reaction [RT-PCR], OR
* Influenza A/H5 cultured from a clinical sample, OR
* High titres (1:80 or higher) of anti-H5 antibodies by microneutralization in convalescent samples of patients who had a compatible illness but no or negative RT-PCR, AND
* The patient survived or if they died an archived biological specimen is available for potential DNA extraction, AND
* Valid, written consent is obtained.
* The biological parents and biological siblings of all the cases and any other family members linking two cases, AND
* Valid, written consent is obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * symptomatic cases with laboratory confirmed H5N1 infection will be eligible for inclusion.
  * Priority for recruitment will be given to cases from multi-case families in order tomaximize the probability of including cases with a genetic etiology.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tawee Chotpitayasunond, Professor, Principal Investigator — Queen Sirikit National Institute of Child Health, Bangkok, Thailand; Herawati Sudoyo, Dr., Principal Investigator — Eijkman Institute for Molecular Biology; Tran Hien Nguyen, Professor, Principal Investigator — National Institute of Hygiene and Epidemiology, Hanoi, Vietnam; Martin Hibberd, Dr., Principal Investigator — Genome Institute of Singapore, Singapore
Locations (1):
- Oxford University Clinical Research Unit, Hanoi, Hanoi, Vietnam

REFERENCES:
- [Background] Albright FS, Orlando P, Pavia AT, Jackson GG, Cannon Albright LA. Evidence for a heritable predisposition to death due to influenza. J Infect Dis. 2008 Jan 1;197(1):18-24. doi: 10.1086/524064. PMID 18171280
- [Background] Apisarnthanarak A, Erb S, Stephenson I, Katz JM, Chittaganpitch M, Sangkitporn S, Kitphati R, Thawatsupha P, Waicharoen S, Pinitchai U, Apisarnthanarak P, Fraser VJ, Mundy LM. Seroprevalence of anti-H5 antibody among Thai health care workers after exposure to avian influenza (H5N1) in a tertiary care center. Clin Infect Dis. 2005 Jan 15;40(2):e16-8. doi: 10.1086/427034. Epub 2004 Dec 17. PMID 15655735
- [Background] Bauer M, Orescovic I, Schoell WM, Bianchi DW, Pertl B. Detection of maternal deoxyribonucleic acid in umbilical cord plasma by using fluorescent polymerase chain reaction amplification of short tandem repeat sequences. Am J Obstet Gynecol. 2002 Jan;186(1):117-20. doi: 10.1067/mob.2002.118306. PMID 11810096
- [Background] Beigel JH, Farrar J, Han AM, Hayden FG, Hyer R, de Jong MD, Lochindarat S, Nguyen TK, Nguyen TH, Tran TH, Nicoll A, Touch S, Yuen KY; Writing Committee of the World Health Organization (WHO) Consultation on Human Influenza A/H5. Avian influenza A (H5N1) infection in humans. N Engl J Med. 2005 Sep 29;353(13):1374-85. doi: 10.1056/NEJMra052211. No abstract available. PMID 16192482
- [Background] Burgner D, Jamieson SE, Blackwell JM. Genetic susceptibility to infectious diseases: big is beautiful, but will bigger be even better? Lancet Infect Dis. 2006 Oct;6(10):653-63. doi: 10.1016/S1473-3099(06)70601-6. PMID 17008174
- [Background] Burton PR, Tobin MD, Hopper JL. Key concepts in genetic epidemiology. Lancet. 2005 Sep 10-16;366(9489):941-51. doi: 10.1016/S0140-6736(05)67322-9. PMID 16154023
- [Background] Buxton Bridges C, Katz JM, Seto WH, Chan PK, Tsang D, Ho W, Mak KH, Lim W, Tam JS, Clarke M, Williams SG, Mounts AW, Bresee JS, Conn LA, Rowe T, Hu-Primmer J, Abernathy RA, Lu X, Cox NJ, Fukuda K. Risk of influenza A (H5N1) infection among health care workers exposed to patients with influenza A (H5N1), Hong Kong. J Infect Dis. 2000 Jan;181(1):344-8. doi: 10.1086/315213. PMID 10608786
- [Background] Chan VS, Chan KY, Chen Y, Poon LL, Cheung AN, Zheng B, Chan KH, Mak W, Ngan HY, Xu X, Screaton G, Tam PK, Austyn JM, Chan LC, Yip SP, Peiris M, Khoo US, Lin CL. Homozygous L-SIGN (CLEC4M) plays a protective role in SARS coronavirus infection. Nat Genet. 2006 Jan;38(1):38-46. doi: 10.1038/ng1698. Epub 2005 Dec 20. PMID 16369534
- [Background] Colhoun HM, McKeigue PM, Davey Smith G. Problems of reporting genetic associations with complex outcomes. Lancet. 2003 Mar 8;361(9360):865-72. doi: 10.1016/s0140-6736(03)12715-8. PMID 12642066
- [Background] Densen P, Weiler JM, Griffiss JM, Hoffmann LG. Familial properdin deficiency and fatal meningococcemia. Correction of the bactericidal defect by vaccination. N Engl J Med. 1987 Apr 9;316(15):922-6. doi: 10.1056/NEJM198704093161506. No abstract available. PMID 3102964
- [Background] Gagneux P, Cheriyan M, Hurtado-Ziola N, van der Linden EC, Anderson D, McClure H, Varki A, Varki NM. Human-specific regulation of alpha 2-6-linked sialic acids. J Biol Chem. 2003 Nov 28;278(48):48245-50. doi: 10.1074/jbc.M309813200. Epub 2003 Sep 18. PMID 14500706
- [Background] Gilsdorf A, Boxall N, Gasimov V, Agayev I, Mammadzade F, Ursu P, Gasimov E, Brown C, Mardel S, Jankovic D, Pimentel G, Ayoub IA, Elassal EM, Salvi C, Legros D, Pessoa da Silva C, Hay A, Andraghetti R, Rodier G, Ganter B. Two clusters of human infection with influenza A/H5N1 virus in the Republic of Azerbaijan, February-March 2006. Euro Surveill. 2006;11(5):122-6. PMID 16757853
- [Background] Glaser L, Conenello G, Paulson J, Palese P. Effective replication of human influenza viruses in mice lacking a major alpha2,6 sialyltransferase. Virus Res. 2007 Jun;126(1-2):9-18. doi: 10.1016/j.virusres.2007.01.011. Epub 2007 Feb 20. PMID 17313986
- [Background] Hamano E, Hijikata M, Itoyama S, Quy T, Phi NC, Long HT, Ha LD, Ban VV, Matsushita I, Yanai H, Kirikae F, Kirikae T, Kuratsuji T, Sasazuki T, Keicho N. Polymorphisms of interferon-inducible genes OAS-1 and MxA associated with SARS in the Vietnamese population. Biochem Biophys Res Commun. 2005 Apr 22;329(4):1234-9. doi: 10.1016/j.bbrc.2005.02.101. PMID 15766558
- [Background] Haralambous E, Dolly SO, Hibberd ML, Litt DJ, Udalova IA, O'dwyer C, Langford PR, Simon Kroll J, Levin M. Factor H, a regulator of complement activity, is a major determinant of meningococcal disease susceptibility in UK Caucasian patients. Scand J Infect Dis. 2006;38(9):764-71. doi: 10.1080/00365540600643203. PMID 16938729
- [Background] He J, Feng D, de Vlas SJ, Wang H, Fontanet A, Zhang P, Plancoulaine S, Tang F, Zhan L, Yang H, Wang T, Richardus JH, Habbema JD, Cao W. Association of SARS susceptibility with single nucleic acid polymorphisms of OAS1 and MxA genes: a case-control study. BMC Infect Dis. 2006 Jul 6;6:106. doi: 10.1186/1471-2334-6-106. PMID 16824203
- [Background] Hibberd ML, Sumiya M, Summerfield JA, Booy R, Levin M. Association of variants of the gene for mannose-binding lectin with susceptibility to meningococcal disease. Meningococcal Research Group. Lancet. 1999 Mar 27;353(9158):1049-53. doi: 10.1016/s0140-6736(98)08350-0. PMID 10199352
- [Background] Hill AV. Aspects of genetic susceptibility to human infectious diseases. Annu Rev Genet. 2006;40:469-86. doi: 10.1146/annurev.genet.40.110405.090546. PMID 17094741
- [Background] Hoebee B, Rietveld E, Bont L, Oosten Mv, Hodemaekers HM, Nagelkerke NJ, Neijens HJ, Kimpen JL, Kimman TG. Association of severe respiratory syncytial virus bronchiolitis with interleukin-4 and interleukin-4 receptor alpha polymorphisms. J Infect Dis. 2003 Jan 1;187(1):2-11. doi: 10.1086/345859. Epub 2002 Dec 13. PMID 12508140
- [Background] Ip WK, Chan KH, Law HK, Tso GH, Kong EK, Wong WH, To YF, Yung RW, Chow EY, Au KL, Chan EY, Lim W, Jensenius JC, Turner MW, Peiris JS, Lau YL. Mannose-binding lectin in severe acute respiratory syndrome coronavirus infection. J Infect Dis. 2005 May 15;191(10):1697-704. doi: 10.1086/429631. Epub 2005 Apr 11. PMID 15838797
- [Background] Janssen R, Bont L, Siezen CL, Hodemaekers HM, Ermers MJ, Doornbos G, van 't Slot R, Wijmenga C, Goeman JJ, Kimpen JL, van Houwelingen HC, Kimman TG, Hoebee B. Genetic susceptibility to respiratory syncytial virus bronchiolitis is predominantly associated with innate immune genes. J Infect Dis. 2007 Sep 15;196(6):826-34. doi: 10.1086/520886. Epub 2007 Aug 10. PMID 17703412
- [Background] Kandun IN, Wibisono H, Sedyaningsih ER, Yusharmen, Hadisoedarsuno W, Purba W, Santoso H, Septiawati C, Tresnaningsih E, Heriyanto B, Yuwono D, Harun S, Soeroso S, Giriputra S, Blair PJ, Jeremijenko A, Kosasih H, Putnam SD, Samaan G, Silitonga M, Chan KH, Poon LL, Lim W, Klimov A, Lindstrom S, Guan Y, Donis R, Katz J, Cox N, Peiris M, Uyeki TM. Three Indonesian clusters of H5N1 virus infection in 2005. N Engl J Med. 2006 Nov 23;355(21):2186-94. doi: 10.1056/NEJMoa060930. PMID 17124016
- [Background] Kash JC, Tumpey TM, Proll SC, Carter V, Perwitasari O, Thomas MJ, Basler CF, Palese P, Taubenberger JK, Garcia-Sastre A, Swayne DE, Katze MG. Genomic analysis of increased host immune and cell death responses induced by 1918 influenza virus. Nature. 2006 Oct 5;443(7111):578-81. doi: 10.1038/nature05181. Epub 2006 Sep 27. PMID 17006449
- [Background] Katz JM, Lim W, Bridges CB, Rowe T, Hu-Primmer J, Lu X, Abernathy RA, Clarke M, Conn L, Kwong H, Lee M, Au G, Ho YY, Mak KH, Cox NJ, Fukuda K. Antibody response in individuals infected with avian influenza A (H5N1) viruses and detection of anti-H5 antibody among household and social contacts. J Infect Dis. 1999 Dec;180(6):1763-70. doi: 10.1086/315137. PMID 10558929
- [Background] Koopmans M, Wilbrink B, Conyn M, Natrop G, van der Nat H, Vennema H, Meijer A, van Steenbergen J, Fouchier R, Osterhaus A, Bosman A. Transmission of H7N7 avian influenza A virus to human beings during a large outbreak in commercial poultry farms in the Netherlands. Lancet. 2004 Feb 21;363(9409):587-93. doi: 10.1016/S0140-6736(04)15589-X. PMID 14987882
- [Background] Kuiken T, Holmes EC, McCauley J, Rimmelzwaan GF, Williams CS, Grenfell BT. Host species barriers to influenza virus infections. Science. 2006 Apr 21;312(5772):394-7. doi: 10.1126/science.1122818. PMID 16627737
- [Background] Kumari K, Gulati S, Smith DF, Gulati U, Cummings RD, Air GM. Receptor binding specificity of recent human H3N2 influenza viruses. Virol J. 2007 May 9;4:42. doi: 10.1186/1743-422X-4-42. PMID 17490484
- [Background] Langhi DM Jr, Bordin JO. Duffy blood group and malaria. Hematology. 2006 Oct;11(5):389-98. doi: 10.1080/10245330500469841. PMID 17607593
- [Background] Liem NT, Lim W; World Health Organization International Avian Influenza Investigation Team, Vietnam. Lack of H5N1 avian influenza transmission to hospital employees, Hanoi, 2004. Emerg Infect Dis. 2005 Feb;11(2):210-5. doi: 10.3201/eid1102.041075. PMID 15752437
- [Background] Lo YM, Lau TK, Chan LY, Leung TN, Chang AM. Quantitative analysis of the bidirectional fetomaternal transfer of nucleated cells and plasma DNA. Clin Chem. 2000 Sep;46(9):1301-9. PMID 10973858
- [Background] Ly S, Van Kerkhove MD, Holl D, Froehlich Y, Vong S. Interaction between humans and poultry, rural Cambodia. Emerg Infect Dis. 2007 Jan;13(1):130-2. doi: 10.3201/eid1301.061014. PMID 17370527
- [Background] Matrosovich MN, Matrosovich TY, Gray T, Roberts NA, Klenk HD. Human and avian influenza viruses target different cell types in cultures of human airway epithelium. Proc Natl Acad Sci U S A. 2004 Mar 30;101(13):4620-4. doi: 10.1073/pnas.0308001101. Epub 2004 Mar 15. PMID 15070767
- [Background] Masuzaki H, Miura K, Miura S, Yoshiura K, Mapendano CK, Nakayama D, Yoshimura S, Niikawa N, Ishimaru T. Labor increases maternal DNA contamination in cord blood. Clin Chem. 2004 Sep;50(9):1709-11. doi: 10.1373/clinchem.2004.036517. No abstract available. PMID 15331519
- [Background] Newport MJ, Huxley CM, Huston S, Hawrylowicz CM, Oostra BA, Williamson R, Levin M. A mutation in the interferon-gamma-receptor gene and susceptibility to mycobacterial infection. N Engl J Med. 1996 Dec 26;335(26):1941-9. doi: 10.1056/NEJM199612263352602. PMID 8960473
- [Background] Nicholls JM, Chan MC, Chan WY, Wong HK, Cheung CY, Kwong DL, Wong MP, Chui WH, Poon LL, Tsao SW, Guan Y, Peiris JS. Tropism of avian influenza A (H5N1) in the upper and lower respiratory tract. Nat Med. 2007 Feb;13(2):147-9. doi: 10.1038/nm1529. Epub 2007 Jan 7. PMID 17206149
- [Background] Olsen SJ, Ungchusak K, Sovann L, Uyeki TM, Dowell SF, Cox NJ, Aldis W, Chunsuttiwat S. Family clustering of avian influenza A (H5N1). Emerg Infect Dis. 2005 Nov;11(11):1799-1801. doi: 10.3201/eid1111.050646. No abstract available. PMID 16422010
- [Background] Oner AF, Bay A, Arslan S, Akdeniz H, Sahin HA, Cesur Y, Epcacan S, Yilmaz N, Deger I, Kizilyildiz B, Karsen H, Ceyhan M. Avian influenza A (H5N1) infection in eastern Turkey in 2006. N Engl J Med. 2006 Nov 23;355(21):2179-85. doi: 10.1056/NEJMoa060601. PMID 17124015
- [Background] Ortiz JR, Katz MA, Mahmoud MN, Ahmed S, Bawa SI, Farnon EC, Sarki MB, Nasidi A, Ado MS, Yahaya AH, Joannis TM, Akpan RS, Vertefeuille J, Achenbach J, Breiman RF, Katz JM, Uyeki TM, Wali SS. Lack of evidence of avian-to-human transmission of avian influenza A (H5N1) virus among poultry workers, Kano, Nigeria, 2006. J Infect Dis. 2007 Dec 1;196(11):1685-91. doi: 10.1086/522158. Epub 2007 Oct 25. PMID 18008254
- [Background] Park AW, Glass K. Dynamic patterns of avian and human influenza in east and southeast Asia. Lancet Infect Dis. 2007 Aug;7(8):543-8. doi: 10.1016/S1473-3099(07)70186-X. PMID 17646027
- [Background] Pitzer VE, Olsen SJ, Bergstrom CT, Dowell SF, Lipsitch M. Little evidence for genetic susceptibility to influenza A (H5N1) from family clustering data. Emerg Infect Dis. 2007 Jul;13(7):1074-6. doi: 10.3201/eid1307.061538. PMID 18214184
- [Background] Price AL, Patterson NJ, Plenge RM, Weinblatt ME, Shadick NA, Reich D. Principal components analysis corrects for stratification in genome-wide association studies. Nat Genet. 2006 Aug;38(8):904-9. doi: 10.1038/ng1847. Epub 2006 Jul 23. PMID 16862161
- [Background] Rimmelzwaan GF, van Riel D, Baars M, Bestebroer TM, van Amerongen G, Fouchier RA, Osterhaus AD, Kuiken T. Influenza A virus (H5N1) infection in cats causes systemic disease with potential novel routes of virus spread within and between hosts. Am J Pathol. 2006 Jan;168(1):176-83; quiz 364. doi: 10.2353/ajpath.2006.050466. PMID 16400021
- [Background] Schultsz C, Dong VC, Chau NV, Le NT, Lim W, Thanh TT, Dolecek C, de Jong MD, Hien TT, Farrar J. Avian influenza H5N1 and healthcare workers. Emerg Infect Dis. 2005 Jul;11(7):1158-9. doi: 10.3201/eid1107.050070. No abstract available. PMID 16032802
- [Background] Sedyaningsih ER, Isfandari S, Setiawaty V, Rifati L, Harun S, Purba W, Imari S, Giriputra S, Blair PJ, Putnam SD, Uyeki TM, Soendoro T. Epidemiology of cases of H5N1 virus infection in Indonesia, July 2005-June 2006. J Infect Dis. 2007 Aug 15;196(4):522-7. doi: 10.1086/519692. Epub 2007 Jun 29. PMID 17624836
- [Background] Shinya K, Ebina M, Yamada S, Ono M, Kasai N, Kawaoka Y. Avian flu: influenza virus receptors in the human airway. Nature. 2006 Mar 23;440(7083):435-6. doi: 10.1038/440435a. PMID 16554799
- [Background] Shioda T, Nakayama EE. Human genetic polymorphisms affecting HIV-1 diseases. Int J Hematol. 2006 Jul;84(1):12-7. doi: 10.1532/IJH97.06100. PMID 16867896
- [Background] Szretter KJ, Gangappa S, Lu X, Smith C, Shieh WJ, Zaki SR, Sambhara S, Tumpey TM, Katz JM. Role of host cytokine responses in the pathogenesis of avian H5N1 influenza viruses in mice. J Virol. 2007 Mar;81(6):2736-44. doi: 10.1128/JVI.02336-06. Epub 2006 Dec 20. PMID 17182684
- [Background] Tecle T, White MR, Crouch EC, Hartshorn KL. Inhibition of influenza viral neuraminidase activity by collectins. Arch Virol. 2007;152(9):1731-42. doi: 10.1007/s00705-007-0983-4. Epub 2007 May 22. PMID 17514488
- [Background] Thanawongnuwech R, Amonsin A, Tantilertcharoen R, Damrongwatanapokin S, Theamboonlers A, Payungporn S, Nanthapornphiphat K, Ratanamungklanon S, Tunak E, Songserm T, Vivatthanavanich V, Lekdumrongsak T, Kesdangsakonwut S, Tunhikorn S, Poovorawan Y. Probable tiger-to-tiger transmission of avian influenza H5N1. Emerg Infect Dis. 2005 May;11(5):699-701. doi: 10.3201/eid1105.050007. PMID 15890122
- [Background] Thorson A, Petzold M, Nguyen TK, Ekdahl K. Is exposure to sick or dead poultry associated with flulike illness?: a population-based study from a rural area in Vietnam with outbreaks of highly pathogenic avian influenza. Arch Intern Med. 2006 Jan 9;166(1):119-23. doi: 10.1001/archinte.166.1.119. PMID 16401820
- [Background] Tran TH, Nguyen TL, Nguyen TD, Luong TS, Pham PM, Nguyen vV, Pham TS, Vo CD, Le TQ, Ngo TT, Dao BK, Le PP, Nguyen TT, Hoang TL, Cao VT, Le TG, Nguyen DT, Le HN, Nguyen KT, Le HS, Le VT, Christiane D, Tran TT, Menno de J, Schultsz C, Cheng P, Lim W, Horby P, Farrar J; World Health Organization International Avian Influenza Investigative Team. Avian influenza A (H5N1) in 10 patients in Vietnam. N Engl J Med. 2004 Mar 18;350(12):1179-88. doi: 10.1056/NEJMoa040419. Epub 2004 Feb 25. PMID 14985470
- [Background] Ungchusak K, Auewarakul P, Dowell SF, Kitphati R, Auwanit W, Puthavathana P, Uiprasertkul M, Boonnak K, Pittayawonganon C, Cox NJ, Zaki SR, Thawatsupha P, Chittaganpitch M, Khontong R, Simmerman JM, Chunsutthiwat S. Probable person-to-person transmission of avian influenza A (H5N1). N Engl J Med. 2005 Jan 27;352(4):333-40. doi: 10.1056/NEJMoa044021. Epub 2005 Jan 24. PMID 15668219
- [Background] van Riel D, Munster VJ, de Wit E, Rimmelzwaan GF, Fouchier RA, Osterhaus AD, Kuiken T. H5N1 Virus Attachment to Lower Respiratory Tract. Science. 2006 Apr 21;312(5772):399. doi: 10.1126/science.1125548. Epub 2006 Mar 23. PMID 16556800
- [Background] Vong S, Coghlan B, Mardy S, Holl D, Seng H, Ly S, Miller MJ, Buchy P, Froehlich Y, Dufourcq JB, Uyeki TM, Lim W, Sok T. Low frequency of poultry-to-human H5NI virus transmission, southern Cambodia, 2005. Emerg Infect Dis. 2006 Oct;12(10):1542-7. doi: 10.3201/eid1210.060424. PMID 17176569
- [Background] Wellcome Trust Case Control Consortium. Genome-wide association study of 14,000 cases of seven common diseases and 3,000 shared controls. Nature. 2007 Jun 7;447(7145):661-78. doi: 10.1038/nature05911. PMID 17554300
- [Background] Yen HL, Lipatov AS, Ilyushina NA, Govorkova EA, Franks J, Yilmaz N, Douglas A, Hay A, Krauss S, Rehg JE, Hoffmann E, Webster RG. Inefficient transmission of H5N1 influenza viruses in a ferret contact model. J Virol. 2007 Jul;81(13):6890-8. doi: 10.1128/JVI.00170-07. Epub 2007 Apr 25. PMID 17459930